CLINICAL TRIAL: NCT03932448
Title: Fever After Tick Bite (FATB) Study; Determining the Etiology of Tick-Borne Human Infections in Northern Europe
Brief Title: Fever After Tick Bite Study
Acronym: FATB
Status: Withdrawn | Type: Observational
Why Stopped: Enrollment in the study was rendered unfeasible due to restrictions and disruptions caused by the COVID-19 pandemic.
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other); Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: FATB Study Group
Record Dates: First submitted 2019-04-16; First posted 2019-04-30 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Tick-Bite; Fever; Tick Fever; Tick-Borne Diseases; Encephalitis, Tick-Borne; Tick Bites
MeSH Terms: conditions — Tick Bites; Fever; Anaplasmosis; Tick-Borne Diseases; Encephalitis, Tick-Borne

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, urine, saliva, and PBMCs will be sampled and stored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: The proposed study is not interventional. — The proposed study is not interventional. However, if a treatable microorganism is detected, e.g. Borrelia or Anaplasma, suitable therapy, e.g. doxycycline, will be in initiated if appropriate.

SUMMARY:
The proposed study is a collaboration between Microbiology, SU/Sahlgrenska and the Infectious Diseases clinic at SU/Östra as well as several Infectious Diseases clinics throughout Sweden aiming at improving microbiological diagnostic assays regarding the early identification of tick-borne microorganisms (including as of yet unidentified pathogens) capable of causing human disease using modern diagnostic tools.

At the initial study visit (day 0) plasma, serum, urine, saliva, and PBMCs (and tick, if available) will be collected from patients developing fever within two weeks after a tick bite. Additional follow-up samples will be obtained after 9 and 30 days as well as after 6 months. The initial samples will be analyzed using (a) directed multiplex PCR analysis for Tick-Borne Encephalitis (TBE), Borrelia, Anaplasma, Neoerlichia, Rickettsia, Coxiella, Tularemia, and Babesiosis in plasma, whole blood and urine, (b) conventional IgM and IgG serology for TBE, (c) "Next Generation Sequencing" (NGS) for the detection of bacterial 16s rRNA as well as unknown viruses, (d) potential biomarkers, and (e) host genetic factors. Among patients where initial sampling indicates the presence of a potential pathogen or in patients developing neurological symptoms, a lumbar puncture will be performed and CSF will be further analyzed. Samples will also be evaluated regarding potential microbiological factors predisposing for severity of infection.

The primary objective of the study is to improve diagnostic tools in the initial early phase of infections caused by tick-borne pathogens, especially TBE prior to the affliction of the central nervous system, and to attempt to identify which factors impact the course of infection as it is believed that approximately 75% of infected individuals resolve their infection in this first phase whereas others develop meningoencephalitis with significant subsequent neurological sequelae. Secondary objectives of the study include investigating for the presence of and treating other tick-borne pathogens, setting the stage for coming clinical trials evaluating novel anti-viral therapies for TBE.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male and female patients ≥18 years of age
* Medical history of tick bite within past 2 weeks
* Documented or medical history of fever (≥38°C) within past 2 weeks

Exclusion Criteria:

* Inability or unwillingness to provide informed consent or abide by the requirements of the study
* Presence of urinary tract symptoms
* Presence of non-tick related, infectious agent causing fever, e.g. a respiratory virus
* Presence of other medical, non-infectious cause of fever

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women ≥18 years old with documented or a medical history of fever (≥38°C) within 2 weeks after a tick bite.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Etiology of fever (≥38°C) developing within 2 weeks after a tick bite. | Up to two weeks after the tick bite.
  Number of participants with detectable Tick-Borne Encephalitis Virus (TBEV), Borrelia, Anaplasma, Neoerlichia, Rickettsia, Coxiella burnetii, Tularemia, and/or Babesia infections.
Proportion of subjects developing neurological symptoms after a tick bite. | Up to six months after the tick bite.
  The proportion of subjects developing neurological symptoms in each of the following etiological categories: Tick-Borne Encephalitis Virus (TBEV), Borrelia, Anaplasma, Neoerlichia, Rickettsia, Coxiella burnetii, Tularemia, and/or Babesia.
Proportion of subjects developing other serious, non-neurological symptoms or disease after a tick bite. | Up to six months after the tick bite.
  The proportion of subjects developing other serious, non-neurological symptoms or disease in each of the following etiological categories: Tick-Borne Encephalitis Virus (TBEV), Borrelia, Anaplasma, Neoerlichia, Rickettsia, Coxiella burnetii, Tularemia, and/or Babesia.

SECONDARY OUTCOMES:
Impact of body mass index (BMI) of subjects on the risk of development of neurological symptoms. | Up to six months after the tick bite.
  Evaluation of body mass index (weight and height will be combined to report BMI in kg/m2) of subjects developing vs. not developing neurological symptoms.
Impact of waist circumference of subjects on the risk of development of neurological symptoms. | Up to six months after the tick bite.
  Evaluation of waist circumference (measured in cm) of subjects developing vs. not developing neurological symptoms.
Impact of gender of subjects on the risk of development of neurological symptoms. | Up to six months after the tick bite.
  Evaluation of gender (male vs. female) of subjects developing vs. not developing neurological symptoms.
Impact of age of subjects on the risk of development of neurological symptoms. | Up to six months after the tick bite.
  Evaluation of age (measured in years) of subjects developing vs. not developing neurological symptoms.
Impact of body mass index of subjects developing other serious, non-neurological symptoms or disease. | Up to six months after the tick bite.
  Evaluation of body mass index (weight and height will be combined to report BMI in kg/m2) of subjects developing vs. not developing other serious, non-neurological symptoms or disease.
Impact of waist circumference of subjects developing other serious, non-neurological symptoms or disease. | Up to six months after the tick bite.
  Evaluation of waist circumference (measured in cm) of subjects developing vs. not developing other serious, non-neurological symptoms or disease.
Impact of gender of subjects developing other serious, non-neurological symptoms or disease. | Up to six months after the tick bite.
  Evaluation of gender (male vs. female) of subjects developing vs. not developing other serious, non-neurological symptoms or disease.
Impact of age of subjects developing other serious, non-neurological symptoms or disease. | Up to six months after the tick bite.
  Evaluation of age (measured in years) of subjects developing vs. not developing other serious, non-neurological symptoms or disease.
Prospective evaluation of the utility of Next Generation Sequencing (NGS) for the detection of unknown viruses and of bacterial 16s rRNA vs. directed Multiplex PCR | Up to 30 days after the tick bite.
  Number of participants with Tick-Borne Encephalitis Virus (TBEV), Borrelia, Anaplasma, Neoerlichia, Rickettsia, Coxiella burnetii, Tularemia, and/or Babesia infections as detected using Next Generation Sequencing (NGS) in comparison to Multiplex Polymerase Chain Reaction (Multiplex PCR).
Prospective evaluation of the specificity and sensitivity of TBEV-RNA and TBE IgM serology in the early phase of infection, i.e. up to 30 days after the tick bite. | Up to 30 days after the tick bite.
  Comparison of the number of subjects correctly identified as being infected with TBEV by means of analysis of TBEV-RNA vs. TBE IgM serology in the early phase of infection, i.e. up to 30 days after the tick bite.
Prospective evaluation of the specificity and sensitivity of TBEV-RNA in urine vs. plasma/whole blood in the early phase of TBE infection, i.e. up to 30 days after the tick bite. | Up to 30 days after the tick bite.
  Comparison of the number of subjects correctly identified as being infected with TBEV by means of analysis of TBEV-RNA in urine vs. plasma/whole blood in the early phase of TBE infection, i.e. up to 30 days after the tick bite.
Prospective evaluation of the specificity and sensitivity of PCR for Borrelia DNA in plasma/serum as well as Borrelia IgM serology in the early phase of infection, i.e. up to 30 days after the tick bite. | Up to 30 days after the tick bite.
  Comparison the number of subjects correctly identified as being infected with Borrelia by means of analysis of PCR for Borrelia DNA in plasma/serum as well as Borrelia IgM and IgG serology in the early phase of infection, i.e. up to 30 days after the tick bite.
Prospective evaluation of the specificity and sensitivity of early evaluation of plasma concentrations of the neurological markers NFL in relation to the likelihood of developing neurological symptoms. | Up to six months after the tick bite.
  Comparison of plasma concentrations of the neurological marker NFL will be evaluated among subjects developing vs. not developing neurological symptoms.
Prospective evaluation of the specificity and sensitivity of early evaluation of plasma concentrations of the neurological marker T-tau in relation to the likelihood of developing neurological symptoms. | Up to six months after the tick bite.
  Comparison of plasma concentrations of the neurological marker T-tau will be evaluated among subjects developing vs. not developing neurological symptoms.
Prospective evaluation of the specificity and sensitivity of early evaluation of plasma concentrations of the neurological marker GFAp in relation to the likelihood of developing neurological symptoms. | Up to six months after the tick bite.
  Comparison of plasma concentrations of neurological marker GFAp will be evaluated among subjects developing vs. not developing neurological symptoms.
Prospective evaluation of the specificity and sensitivity of early evaluation of plasma concentrations of IP-10 (aka CXCL10) in relation to the likelihood of developing neurological symptoms. | Up to six months after the tick bite.
  Comparison of plasma concentrations of IP-10 (aka CXCL10) will be evaluated among subjects developing vs. not developing neurological symptoms.
Prospective evaluation of the specificity and sensitivity of early evaluation of 25-hydroxy vitamin D (25(OH)D) concentrations in relation to the likelihood of developing neurological symptoms. | Up to six months after the tick bite.
  Comparison of plasma concentrations of 25-hydroxy vitamin D (25(OH)D) will be evaluated among subjects developing vs. not developing neurological symptoms.
Prospective evaluation of peripheral blood mononuclear cells (PBMCs) analyzed by FACS, in relation to the likelihood of developing neurological symptoms. | Up to six months after the tick bite.
  Comparison of the proportion of CD56 negative NK, CD4+ CD38+, CD8+ CD38+, CD8+CD16+, Foxp3+, and pDC (CD303+) cells analyzed by FACS will be evaluated among subjects developing vs. not developing neurological symptoms.
Prospective evaluation of the impact of host genetic polymorphisms in the IFNL4 gene in relation to the likelihood of developing neurological symptoms. | Up to six months after the tick bite.
  Proportion of subjects with genetic polymorphisms in the IFNL4 gene evaluated among subjects developing vs. not developing neurological symptoms.
Prospective evaluation of the impact of host genetic polymorphisms in the ITPA gene in relation to the likelihood of developing neurological symptoms. | Up to six months after the tick bite.
  Proportion of subjects with genetic polymorphisms in the ITPA gene evaluated among subjects developing vs. not developing neurological symptoms.
Prospective evaluation of the impact of prior vaccination against TBE on frequency and outcome of TBEV infection. | From time of prior vaccination until six months after the tick bite.
  Comparison of subjects with vs. without prior vaccination against TBE on frequency and outcome of TBEV infection.
Prospective evaluation of the impact of prior vaccination against Yellow Fever on frequency and outcome of TBEV infection. | From time of prior vaccination until six months after the tick bite.
  Comparison of subjects with vs. without prior vaccination against Yellow Fever on frequency and outcome of TBEV infection.
Prospective evaluation of the impact of prior vaccination against Japanese Encephalitis on frequency and outcome of TBEV infection. | From time of prior vaccination until six months after the tick bite.
  Comparison of subjects with vs. without prior vaccination against Japanese Encephalitis on frequency and outcome of TBEV infection.
Prospective evaluation of the association between presence or absence of immunosuppression in relation to the likelihood of developing neurological symptoms. | Up to six months after the tick bite.
  The proportion of subjects with vs. without immunosuppression will be evaluated among subjects developing vs. not developing neurological symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Lagging, MD, PhD, Principal Investigator — Göteborg University
Locations (1):
- Dept. of Infectious Diseases, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided